CLINICAL TRIAL: NCT07074483
Title: Accuracy of AuReha for Measuring Upper Limb Movements Compared to "Usual Care"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DigitalRehab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DigitalRehab_01_2024
Record Dates: First submitted 2025-06-11; First posted 2025-07-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: measurement accuracy; wearable medical device; inertial measurement sensors; upper limb rehabilitation; monitoring system; supporting system; Rehabilitation technology validation; Goniometer comparison
MeSH Terms: interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers participants (Experimental): This arm includes healthy adult volunteers who will perform a series of upper limb rehabilitation exercises using the AuReha system, as the aim of the study is to evaluate the accuracy of the device in capturing upper limb joint movements, as well as to assess the usability and user experience of the wearable system.
  No therapeutic or diagnostic interventions will be administered, as this is a non-invasive study focused on system validation and user feedback.
  Interventions: Device: Upper limb rehabilitation wearable device

INTERVENTIONS:
Device: Upper limb rehabilitation wearable device — The intervention consists in using the AuReha system to perform a series of upper limb rehabilitation exercises.
  No therapeutic or diagnostic interventions will be administered, as this is a non-invasive study focused on system validation and user feedback.
  Other Names: sensorized garment; wearable device for upper limb data detection

SUMMARY:
The clinical investigation design involves a validation study conducted on a group of healthy volunteers.

It is an interventional, monocentric study with a paired data design, aimed at verifying the equivalence of the AuReha system compared to the usual care system (goniometer) in the measurement of biomechanical parameters.

In addition to the measurements taken with AuReha and the goniometer, additional data collection will be carried out using the Kinovea system, which involves video analysis of recorded movement and has demonstrated high accuracy.

The validation on healthy volunteers will be conducted at the Laboratory of Movement and Sport Science (LaMSS) of the IRCCS Ospedale Galeazzi-Sant'Ambrogio in Milan, and will include the recruitment of 96 volunteers from among the hospital's internal staff.

DETAILED DESCRIPTION:
The primary objective of the clinical investigation is to obtain CE certification for the device.

Specifically, the project aims to document the accuracy of motion measurements detected by AuReha by comparing them with the most commonly used system in current "usual care" for upper limb rehabilitation: the goniometer. At the same time, the investigation will assess the correct and timely transmission of data collected by the AuReha device within the standalone software platform, which is composed of two main functional modules: one for the subject/patient and one for healthcare professionals.

These are the foundations for the optimal management of the rehabilitation process, resulting in a system capable of guiding the patient through the proper execution of rehabilitation movements as prescribed by the physician, while also collecting biomechanical parameters for close monitoring of the patient's response to the therapy.

In addition to the goal of certifying the AuReha system through evidence of motion measurement accuracy, the study will also include descriptive evaluations/objectives related to user experience and the usability/wearability of the smart shirt.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Volunteers who provide written informed consent to participate in the study
* Absence of movement limitations affecting the upper limbs and/or trunk

Exclusion Criteria:

* Pregnant and/or breastfeeding women (verified through self-declaration)
* Epilepsy
* Allergy or hypersensitivity to materials used in the medical device, specifically: polypropylene and lycra (fabric), nylon (integrated zipper), viscose and elastane (zipper integration fabric)
* Chronic headache under treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The equivalence of AuReha compared to "Usual Care" (goniometer-based system) in measuring the shoulder's medio-lateral range of motion angle (abduction). | Day 1
  The shoulder joint, also known as the glenohumeral joint, is a ball-and-socket type articulation formed by the head of the humerus and the glenoid cavity of the scapula. Flexion and extension are movements that occur around the coronal axis.
  Abduction and adduction are movements that occur around the sagittal axis. Abduction is a lateral movement ranging from 0° (arm perpendicular to the floor) to a vertical position above the head (approximately 180°).
  This final position is equivalent to that reached during flexion and involves the coordinated movement of the shoulder girdle and the glenohumeral joint.

SECONDARY OUTCOMES:
Equivalence in the measurement of the shoulder and elbow flexion ranges of motion | Day 1
  The equivalence of the measurements derived from AuReha and the instrument of comparison will be measured in degrees.
  The elbow is a hinge joint formed by the articulation of the humerus with the ulna and radius. Flexion and extension occur along a coronal axis and are the two primary movements allowed by this joint. Flexion is an anterior movement that ranges from a fully extended position (0 degrees) to full flexion (approximately 145°).
  Shoulder flexion is an anterior movement with a range starting from the anatomical position of 0° (arm perpendicular to the ground) up to 180° overhead. However, this final position is achieved only through a combination of movements involving both the shoulder joint and the shoulder girdle. The glenohumeral joint alone can flex to approximately 120°, while the remaining 60° are achieved through scapular abduction and lateral rotation, which reorients the glenoid cavity and allows the humerus to reach a fully vertical position.
Characterization of AuReha in measuring movement smoothness and its timely and accurate transmission to the therapists' platform | Day 1
  "Movement Smoothness" is a parameter calculated by the AuRhea Web Platform and it evaluates the continuity and coordination of performed movements. It is measured through jerk, which refers to the variation in movement velocity.
  Unit of Measure: Percentage (%)
  The accuracy and timeliness of this parameter transfers to the AuReha Web Platform will be assessed by verifying that is registered on the platform in real time, immediately upon detection by the AuReha Sensorized Shirt.
Characterization of AuReha in measuring movement accuracy and its timely and accurate transmission to the therapists' platform | Day 1
  "Movement accuracy" is a parameter calculated by the AuRhea Web Platform and it measures how precisely the volunteer performs the prescribed movements by comparing the deviation of the executed trajectory from the ideal one.
  Unit of Measure: Percentage (%)
  The accuracy and timeliness of this parameter transfers to the AuReha Web Platform will be assessed by verifying that is registered on the platform in real time, immediately upon detection by the AuReha Sensorized Shirt.
Characterization of AuReha in measuring trunk stability and its timely and accurate transmission to the therapists' platform | Day 1
  "Trunk stability" is a parameter calculated by the AuRhea Web Platform and it assesses the inclination of the trunk across the three reference planes (frontal, sagittal, and transverse) during the execution of exercises.
  Unit of Measure: Percentage (%)
  The accuracy and timeliness of this parameter transfers to the AuReha Web Platform will be assessed by verifying that is registered on the platform in real time, immediately upon detection by the AuReha Sensorized Shirt.
Characterization of AuReha in measuring limb compensation and its timely and accurate transmission to the therapists' platform | Day 1
  "Limb compensation" is a parameter calculated by the AuRhea Web Platform and it monitors any incorrect compensatory movements performed by the limbs during exercises.
  Unit of Measure: Percentage (%)
  The accuracy and timeliness of this parameter transfers to the AuReha Web Platform will be assessed by verifying that is registered on the platform in real time, immediately upon detection by the AuReha Sensorized Shirt.
Characterization of AuReha in measuring the percentage of correct movements executed by the subject, and its timely and accurate transmission to the therapists' platform | Day 1
  "Percentage of correct movements" is a parameter calculated by the AuRhea Web Platform and it indicates the percentage of movements correctly performed by the volunteer in relation to the total number of goals proposed in the session. The number of proposed goals in each section varies based on the volunteer's performance, thanks to an adaptive algorithm.
  Unit of Measure: Percentage (%)
  The accuracy and timeliness of this parameter transfers to the AuReha Web Platform will be assessed by verifying that is registered on the platform in real time, immediately upon detection by the AuReha Sensorized Shirt.
Correlation between AuReha shirt size (categorical: XS, S, M, L,) and the anthropometric measurements of healthy volunteers (in cm) | Day 1
  Evaluation of AuReha's fit on healthy volunteers, through the assessment of the correlation between the selected shirt size (categorical: XS, S, M, L) and continuous anthropometric variables, including body circumferences and segment lengths. Circumferences (in cm) will include: chest, waist, hips, upper arm, and forearm. Segment lengths (in cm) will include: shoulder to iliac spine and shoulder to wrist. All measurements will be taken using a standard anthropometric tape measure.
Characterization of AuReha in terms of usability for healthy volunteers | Day 1
  Assessment of the usability of AuReha by healthy volunteers. Custom questionnaires developed for this purpose are annexed to the clinical protocol. In particular, the questionnaire collects user feedback on the AuReha App and sensorized shirt, focusing on usability, instruction clarity, and garment fit. It combines Yes/No items, a 0-4 Likert difficulty scale (from "no difficulty" to "system unusable"), and open-text fields for qualitative insights.
Characterization of AuReha in terms of usability for healthcare professionals | Day 1
  Assessment of the usability of AuReha by healthcare professionals. Custom questionnaires developed for this purpose are annexed to the clinical protocol. In particular, the surveys gauge healthcare professionals' experience with the AuReha Web Platform, assessing data transfer reliability, information clarity, user satisfaction, and decision-support effectiveness. It combines yes/no questions with open-text fields for detailed feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi - Sant'Ambrogio, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided